CLINICAL TRIAL: NCT04005404
Title: Surgical Treatment of Proximal Femoral Fractures Under Peripheral Regional Anesthesia. A Prospective Pilot Study
Brief Title: Surgical Treatment of Hip Fractures Under Peripheral Regional Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Research Center (Other)
Responsible Party: Principal Investigator, Dr.med.Ronald Seidel, Principal Investigator, Helios Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A 2018 0237
Record Dates: First submitted 2019-06-29; First posted 2019-07-02 (Actual); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hip Fractures
Keywords: Regional Anesthesia; Ultrasonography; Hip Fractures; Lumbosacral Plexus
MeSH Terms: conditions — Hip Fractures | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Differentiated analysis for the subgroups "subtrochanteric femoral fractures", "intertrochanteric femoral fractures" and "neck femur fractures"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intertrochanteric femoral fractures (Experimental): geriatric patients with intertrochanteric femoral fracture who have consented to the study intervention
  Interventions: Drug: Ropivacaine (sciatic nerve block); Drug: Ropivacaine (lumbar plexus block L2-L4); Drug: Ropivacaine (lumbar plexus block Th12-L1)
- neck femur fractures (Experimental): geriatric patients with neck of femur fracture who have consented to the study intervention
  Interventions: Drug: Ropivacaine (sciatic nerve block); Drug: Ropivacaine (lumbar plexus block L2-L4); Drug: Ropivacaine (lumbar plexus block Th12-L1)
- subtrochanteric femoral fractures (Experimental): geriatric patients with subtrochanteric femoral fracture who have consented to the study intervention
  Interventions: Drug: Ropivacaine (sciatic nerve block); Drug: Ropivacaine (lumbar plexus block L2-L4); Drug: Ropivacaine (lumbar plexus block Th12-L1)

INTERVENTIONS:
Drug: Ropivacaine (sciatic nerve block) — injection of 20 ml ropivacaine 0.375%
  Other Names: parasacral sciatic nerve block (sacral plexus)
Drug: Ropivacaine (lumbar plexus block L2-L4) — injection of 20 ml ropivacaine 0.375%
  Other Names: posts compartment block (lumbar plexus L2-L4)
Drug: Ropivacaine (lumbar plexus block Th12-L1) — injection of 20 ml ropivacaine 0.375%
  Other Names: transmuscular quadratus lumborum block (lumbar plexus Th12-L1)

SUMMARY:
The study investigates whether treatment of proximal femoral fractures is possible using a peripheral regional anesthesia technique.

DETAILED DESCRIPTION:
The study investigates whether treatment of proximal femoral fractures is possible using a peripheral regional anesthesia technique.

After positioning on the non-fractured side, a double injection technique is used (dual guidance concept: nerve stimulation and sonography).

The injections are performed parasacrally (blockade of the sacral plexus under the piriformis muscle) and lumbar paravertebrally (psoas compartment block and transmuscular quadratus lumborum block). Per block 20 ml ropivacaine 0.375% is administered (total dose: 225mg ropivacaine).

The study examines the success rate (rate of successfully performed nerve blockade; need for supplemental medication: sufentanil and/or propofol; conversion rate to general anesthesia), circulatory stability (need for application of ephedrine or norepinephrine) and side effects.

ELIGIBILITY:
Inclusion Criteria:

* proximal femoral fracture
* older then 18 years
* written informed consent

Exclusion Criteria:

* local or systematic inflammation
* allergy to ropivacaine
* participate in other studies
* body mass index over 35
* periprosthetic fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Helios Medical Center Schwerin, Department of Anesthesiology, Schwerin, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikary SD, Short AJ, El-Boghdadly K, Abdelmalak MJ, Chin KJ. Transmuscular quadratus lumborum versus lumbar plexus block for total hip arthroplasty: A retrospective propensity score matched cohort study. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):372-378. doi: 10.4103/joacp.JOACP_335_17. PMID 30386022
- [Background] Akkaya T, Comert A, Kendir S, Acar HI, Gumus H, Tekdemir I, Elhan A. Detailed anatomy of accessory obturator nerve blockade. Minerva Anestesiol. 2008 Apr;74(4):119-22. PMID 18354367
- [Background] Birnbaum K, Prescher A, Hessler S, Heller KD. The sensory innervation of the hip joint--an anatomical study. Surg Radiol Anat. 1997;19(6):371-5. doi: 10.1007/BF01628504. PMID 9479711
- [Background] Coburn M, Sanders RD, Maze M, Nguyen-Pascal ML, Rex S, Garrigues B, Carbonell JA, Garcia-Perez ML, Stevanovic A, Kienbaum P, Neukirchen M, Schaefer MS, Borghi B, van Oven H, Tognu A, Al Tmimi L, Eyrolle L, Langeron O, Capdevila X, Arnold GM, Schaller M, Rossaint R; HIPELD Study Investigators. The hip fracture surgery in elderly patients (HIPELD) study to evaluate xenon anaesthesia for the prevention of postoperative delirium: a multicentre, randomized clinical trial. Br J Anaesth. 2018 Jan;120(1):127-137. doi: 10.1016/j.bja.2017.11.015. Epub 2017 Nov 21. PMID 29397119
- [Background] Duan X, Coburn M, Rossaint R, Sanders RD, Waesberghe JV, Kowark A. Efficacy of perioperative dexmedetomidine on postoperative delirium: systematic review and meta-analysis with trial sequential analysis of randomised controlled trials. Br J Anaesth. 2018 Aug;121(2):384-397. doi: 10.1016/j.bja.2018.04.046. Epub 2018 Jun 22. PMID 30032877
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Guay J, Parker MJ, Gajendragadkar PR, Kopp S. Anaesthesia for hip fracture surgery in adults. Cochrane Database Syst Rev. 2016 Feb 22;2(2):CD000521. doi: 10.1002/14651858.CD000521.pub3. PMID 26899415
- [Background] Guay J, Parker MJ, Griffiths R, Kopp SL. Peripheral Nerve Blocks for Hip Fractures: A Cochrane Review. Anesth Analg. 2018 May;126(5):1695-1704. doi: 10.1213/ANE.0000000000002489. PMID 28991122
- [Background] Johnston DF, Stafford M, McKinney M, Deyermond R, Dane K. Peripheral nerve blocks with sedation using propofol and alfentanil target-controlled infusion for hip fracture surgery: a review of 6 years in use. J Clin Anesth. 2016 Mar;29:33-9. doi: 10.1016/j.jclinane.2015.10.012. Epub 2016 Feb 2. PMID 26897445
- [Background] Nielsen TD, Moriggl B, Soballe K, Kolsen-Petersen JA, Borglum J, Bendtsen TF. A Cadaveric Study of Ultrasound-Guided Subpectineal Injectate Spread Around the Obturator Nerve and Its Hip Articular Branches. Reg Anesth Pain Med. 2017 May/Jun;42(3):357-361. doi: 10.1097/AAP.0000000000000587. PMID 28263244
- [Background] Sa M, Graca R, Reis H, Cardoso JM, Sampaio J, Pinheiro C, Machado D. [Superior gluteal nerve: a new block on the block?]. Braz J Anesthesiol. 2018 Jul-Aug;68(4):400-403. doi: 10.1016/j.bjan.2016.11.001. Epub 2017 May 24. PMID 28551063
- [Background] Sauter AR, Ullensvang K, Niemi G, Lorentzen HT, Bendtsen TF, Borglum J, Pripp AH, Romundstad L. The Shamrock lumbar plexus block: A dose-finding study. Eur J Anaesthesiol. 2015 Nov;32(11):764-70. doi: 10.1097/EJA.0000000000000265. PMID 26426575
- [Background] Short AJ, Barnett JJG, Gofeld M, Baig E, Lam K, Agur AMR, Peng PWH. Anatomic Study of Innervation of the Anterior Hip Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 Feb;43(2):186-192. doi: 10.1097/AAP.0000000000000701. PMID 29140962
- [Background] Taha AM. A simple and successful sonographic technique to identify the sciatic nerve in the parasacral area. Can J Anaesth. 2012 Mar;59(3):263-7. doi: 10.1007/s12630-011-9630-3. Epub 2011 Dec 3. PMID 22139964
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Van Waesberghe J, Stevanovic A, Rossaint R, Coburn M. General vs. neuraxial anaesthesia in hip fracture patients: a systematic review and meta-analysis. BMC Anesthesiol. 2017 Jun 28;17(1):87. doi: 10.1186/s12871-017-0380-9. PMID 28659127
- [Background] White SM, Moppett IK, Griffiths R, Johansen A, Wakeman R, Boulton C, Plant F, Williams A, Pappenheim K, Majeed A, Currie CT, Grocott MP. Secondary analysis of outcomes after 11,085 hip fracture operations from the prospective UK Anaesthesia Sprint Audit of Practice (ASAP-2). Anaesthesia. 2016 May;71(5):506-14. doi: 10.1111/anae.13415. Epub 2016 Mar 4. PMID 26940645

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intertrochanteric Femoral Fractures | Neck Femur Fractures | Subtrochanteric Femoral Fractures
Started | 43 | 34 | 3
Completed | 42 | 33 | 3
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intertrochanteric Femoral Fractures | Neck Femur Fractures | Subtrochanteric Femoral Fractures | Total
Number analyzed (Participants) | 42 | 33 | 3 | 78
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 87 [81.75 to 89.25] | 84 [80.5 to 87] | 79 [72 to 91] | 85 [81 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 19 | 3 | 53
  Male | 11 | 14 | 0 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 42 | 33 | 3 | 78
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 42 | 33 | 3 | 78

OUTCOME MEASURES:

1. Primary Outcome: Success Rate (Supplemental Medication)
Description: number of participants with need for supplemental analgesic medication (sufentanil)
Time Frame: during surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intertrochanteric Femoral Fractures | Neck Femur Fractures | Subtrochanteric Femoral Fractures
Number analyzed (Participants) | 42 | 33 | 3
Participants | 22 | 20 | 3

2. Primary Outcome: Success Rate (Conversion to General Anesthesia)
Description: number of participants with need for conversion to general anesthesia
Time Frame: during surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intertrochanteric Femoral Fractures | Neck Femur Fractures | Subtrochanteric Femoral Fractures
Number analyzed (Participants) | 42 | 33 | 3
Participants | 1 | 3 | 1

3. Secondary Outcome: Circulation Stability
Description: number of participants with need for application of ephedrine and/or norepinephrine
Time Frame: during surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intertrochanteric Femoral Fractures | Neck Femur Fractures | Subtrochanteric Femoral Fractures
Number analyzed (Participants) | 42 | 33 | 3
Participants | 15 | 15 | 2

ADVERSE EVENTS:
Time Frame: 30 days after surgery
Arm/Group | Intertrochanteric Femoral Fractures | Neck Femur Fractures | Subtrochanteric Femoral Fractures
All-Cause Mortality (participants affected / at risk) | 6/42 | 3/33 | 0/3
Serious Adverse Events (participants affected / at risk) | 21/42 | 16/33 | 0/3
Other Adverse Events (participants affected / at risk) | 0/42 | 0/33 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intertrochanteric Femoral Fractures (N=42) | Neck Femur Fractures (N=33) | Subtrochanteric Femoral Fractures (N=3)
epidural anesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — unintentional epidural anesthesia after lumbar plexus block
delirium (Nervous system disorders) | 5 (5) | 3 (3) | 0 (0) — postoperative delirium
kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0) — acute or acute-on-chronic kidney injury
ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — ventricular tachycardia
heart failure (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) — heart failure
myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) — myocardial infarction
urinary tract infection (Renal and urinary disorders) | 4 (4) | 2 (2) | 0 (0) — urinary tract infection
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) — Pneumonia
hematoma (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
wound infection (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT04005404/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT04005404/SAP_001.pdf